CLINICAL TRIAL: NCT05968625
Title: Post-Treatment Stability, Changes in Mechanical Properties and Patients' OHRQoL Of Direct 3D-Printed Retainers Versus Thermoformed Retainers: An Open-label Randomized Controlled Trial
Brief Title: 3D-Printed Vs Thermoformed Retainers: Comparison of Post-Treatment Stability, Changes in Mechanical Properties and Patients' OHRQoL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, DR BOO HUI SHAN, Principle Investigator, Doctorate (Orthodontics) Postgraduate Student, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: UNIVERSITI MALAYA; UMG013E-2023 (Other Grant/Funding Number: UNIVERSITY GRANT, UNIVERSITI MALAYA)
Record Dates: First submitted 2023-07-17; First posted 2023-08-01 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Orthodontic Retention
Keywords: Thermoformed retainers; 3D-printed retainers; vacuum-formed retainers; Post-treatment stability; Orthodontics

STUDY DESIGN:
Intervention Model Description: Direct 3D-printed retainers
Who Masked: Outcomes Assessor
Masking Description: This is a single-blinded study, where the statistician that analyzes the data is blinded. The subjects are impossible to blind due to subtle differences in the physical appearance of both appliances.
  Blinding of the operator will not be possible due to the differences in clinical procedures involved in fabrication of TFR and 3DPR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermoformed retainers (TFR) (Experimental): Thermoformed retainers are constructed from an Erkodur blank (ERKODENT® Erich Kopp GmbH, Pfalzgrafenweiler, Germany) with 1.0 mm in thickness, following the manufacturer's instructions.
  Interventions: Device: Thermoformed retainers
- Direct 3-D printed retainers (3DPR) (Experimental): Private dental laboratories directly print the retainers using a NextDent 3D printer and NextDent ortho Flex resin. Thickness of 0.80mm
  Interventions: Device: 3D-printed retainers

INTERVENTIONS:
Device: Thermoformed retainers — conventional thermoformed retainers fabricated on stone models.
  Arms: Thermoformed retainers (TFR)
Device: 3D-printed retainers — 3D-printed retainers fabricated directly by DLP printer.
  Arms: Direct 3-D printed retainers (3DPR)

SUMMARY:
Following completion of orthodontic treatment, prolonged retention with either part-time or full-time wear of retainers is crucial in preventing relapse. Clear thermoformed retainers (TFR) are easy to fabricate and popular among orthodontic patients. With the advent of digital orthodontics and the development of biocompatible photopolymerizable resin, it is now possible to fabricate direct 3D-printed retainers.

The aim of this study is to determine and compare the post-treatment stability of dentition, changes in thickness and mechanical properties of the retainers, and oral health-related quality of life (OHRQoL) of patients wearing direct 3D-printed retainers and conventional thermoformed retainers over a retention period of 6 months.

DETAILED DESCRIPTION:
Primary Objective:

1. To determine and compare the post-treatment stability for direct 3D printed retainers (3DPR) and conventional TFR (TFR) at baseline (T0), 3 months (T1) and 6 months (T2).

Secondary Objectives:

1. To determine and compare the thickness and mechanical properties for 3DPR and TFR after 6 months of usage.
2. To determine and compare the OHRQoL of patients wearing 3DPR and TFR at T0, T1 and T2.

Sample size calculation:

Sample size calculation is based on the study done by Kumar & Bansal (2011) which compared the effectiveness of two different removable retainers on stability. With an effect size of 1.127, α = 0.05, and power = 0.80. Using G*Power version 3.1.9.7 software, the total number of samples is n = 22 (11 subject per group). This number is increased by 30% to account for the dropout rate to produce the final sample size, n = 30 (15 subjects per group).

Methodology:

Subjects who have completed their orthodontic treatment (fulfil the inclusion and exclusion criteria) and are ready for debond, will be invited to participate in the research and consecutively recruited, between April 2023 until September 2023, in the Postgraduate Orthodontic Clinic, Dental Specialists and Research Tower, Faculty of Dentistry, Universiti Malaya, Malaysia. Patient information sheets and consent forms will be issued to the subjects that fulfil the criteria. Only consented respondents will be recruited.

All 30 subjects will be randomly allocated (simple randomization with 1:1 allocation) to either the TFR group or the 3DPR group by using number generated list provided by www.random.org . The randomization will be performed by the main supervisor, who is not involve in the treatment, data collection and data analysis of the research. The operator will be concealed from the group allocation. The allocation will be revealed to the operator on the day of debond appointment with a opaque white envelope.

All the subjects will undergo the same standard debond process. and receive a post debond thermoformed retainers within 24 hours which they are required to part-time for every night (8-12 hours).

The subjects will be reviewed after 1 week (T0) for scanning of teeth with Trios 3 intraoral scanner. The interventional retainers (TFR or 3DPR) will be issued after 2 weeks. The subjects are instructed to wear the retainers part-time (8-12 hours) for every nights. A pamphlet that contains detailed information on the care of retainers will also be provided to every subject. All the subjects will be reviewed after 3 months (T1) and at 6 months (T2) after wearing the interventional retainers.

The primary outcome is to assess the post-treatment stability after part time wear of the retainers for a period of 6 months. The subject's upper and lower dentition will be scanned by using intraoral scanner at T0, T1, and T2. The measurements will be performed digitally using 3Shape orthodontic analyzer software. Overjet, overbite, intermolar width, and little irregularity index will be measured.

OHIP-14 questionnaire will be given to the participants to answer during T0, T1 and T2. All the retainers will be retrieved at T2 to undergo mechanical test.

Statistical Analysis:

The data collected will be entered into SPSS software (version 26.0). i. Chi-square tests will be used to compare baseline characteristics between the 2 groups.

ii. Repeated measures ANOVA or paired t-test will be used to determine the mean differences in post treatment stability, thickness of retainers, mechanical properties of retainers and OHIP-14 scores at different time intervals. The p-value will be set to less than 0.05.

iii. Two samples independent t test will be used to compare the post-treatment stability, changes in thickness, mechanical properties, and OHIP-14 scores between TFR and 3DPR group. The p-value will be set to less than 0.05.

iv. Shapiro-Wilk tests will be referred, and non-parametric tests will be performed for skewed data.

Data will be analyzed following the intention-to-treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Fixed appliance treatment in both arches and indicated for VFR in the retention phase as part of their original treatment plan.
* No intention to relocate within the study period; able to attend the three-monthly review appointments for half a year.

Exclusion Criteria:

* Single-arch or sectional fixed appliances.
* Space dentition.
* Hypodontia requiring tooth replacement on the retainer as a temporary measure.
* Previous treatment with maxillary expansion.
* Indicated for fixed retainer or double retention regime (such as VFRs fitted over fixed retainers).
* Premature debond from the original fixed appliances course.
* Cleft lip and/or palate; or orthognathic cases.
* Learning difficulties and inability to read written instructions/ questionnaire in English or Malay

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Post-treatment stability | 6 months
  The subject's upper and lower dentition will be scanned by using intraoral scanner at T0, T1, and T2. The measurements will be performed digitally using 3Shape orthodontic Analyzer software (3Shape A/S, Copenhagen, Denmark). Measurements: Overjet (mm), Overbite (mm), Intermolar width (mm), and little irregularity index (mm). All the measurements are in millimetres.

SECONDARY OUTCOMES:
Changes in thickness of retainers | 6 months
  Measurements of changes in thickness (mm) will be performed by the principal investigator by using an electronic digital thickness gauge with a resolution of 0.01 mm and accuracy of ±0.02 mm, which will be calibrated before each use.
Changes in hardness of retainers | 6 months
  The extra sets of retainers (5 sets from each group) at T0 and the retrieved retainers (5 sets from each group) at T2 of each group will be tested. The hardness that will be determined is Vickers hardness in Megapascal (MPa). A universal hardness testing machine (DUH-211S, Shimadzu, Kyoto Japan) will be used to determine the hardness.
Oral Health Impact Profile -14 (OHIP-14) | 6 months
  This research will use the validated Modified short version of the OHIP-14 for Malaysian adults with questions that are relevant to subjects wearing removable retainers. Responses to each item will be scored on a five-point Likert scale measuring from never (score 0) to very often (score 4). The OHIP-14 questionnaire will be given to the participants to answer during T0, T1 and T2.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Dr. Saritha Sivarajan, Study Director — Faculty of Dentistry, Universiti Malaya
Locations (1):
- Orthodontic Postgraduate Clinic, Faculty of Dentistry, Universiti Malaya., Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams A, Bencharit S, Yang IH, Stilianoudakis SC, Carrico CK, Tufekci E. Effect of print angulation on the accuracy and precision of 3D-printed orthodontic retainers. Am J Orthod Dentofacial Orthop. 2022 Jan;161(1):133-139. doi: 10.1016/j.ajodo.2021.01.020. PMID 35012743
- [Background] Rowland H, Hichens L, Williams A, Hills D, Killingback N, Ewings P, Clark S, Ireland AJ, Sandy JR. The effectiveness of Hawley and vacuum-formed retainers: a single-center randomized controlled trial. Am J Orthod Dentofacial Orthop. 2007 Dec;132(6):730-7. doi: 10.1016/j.ajodo.2006.06.019. PMID 18068589
- [Background] Naeem OA, Bencharit S, Yang IH, Stilianoudakis SC, Carrico C, Tufekci E. Comparison of 3-dimensional printing technologies on the precision, trueness, and accuracy of printed retainers. Am J Orthod Dentofacial Orthop. 2022 Apr;161(4):582-591. doi: 10.1016/j.ajodo.2021.03.016. PMID 35337648
- [Background] Kumar AG, Bansal A. Effectiveness and acceptability of Essix and Begg retainers: a prospective study. Aust Orthod J. 2011 May;27(1):52-6. PMID 21696115
- [Background] Kessler A, Hickel R, Reymus M. 3D Printing in Dentistry-State of the Art. Oper Dent. 2020 Jan/Feb;45(1):30-40. doi: 10.2341/18-229-L. Epub 2019 Jun 7. PMID 31172871
- [Background] Jindal P, Juneja M, Siena FL, Bajaj D, Breedon P. Mechanical and geometric properties of thermoformed and 3D printed clear dental aligners. Am J Orthod Dentofacial Orthop. 2019 Nov;156(5):694-701. doi: 10.1016/j.ajodo.2019.05.012. PMID 31677678
- [Background] Etemad-Shahidi Y, Qallandar OB, Evenden J, Alifui-Segbaya F, Ahmed KE. Accuracy of 3-Dimensionally Printed Full-Arch Dental Models: A Systematic Review. J Clin Med. 2020 Oct 20;9(10):3357. doi: 10.3390/jcm9103357. PMID 33092047
- [Background] Cousley RR. Introducing 3D printing in your orthodontic practice. J Orthod. 2020 Sep;47(3):265-272. doi: 10.1177/1465312520936704. Epub 2020 Jul 6. PMID 32627658
- [Background] Cole D, Bencharit S, Carrico CK, Arias A, Tufekci E. Evaluation of fit for 3D-printed retainers compared with thermoform retainers. Am J Orthod Dentofacial Orthop. 2019 Apr;155(4):592-599. doi: 10.1016/j.ajodo.2018.09.011. PMID 30935614
- [Background] Can E, Panayi N, Polychronis G, Papageorgiou SN, Zinelis S, Eliades G, Eliades T. In-house 3D-printed aligners: effect of in vivo ageing on mechanical properties. Eur J Orthod. 2022 Jan 25;44(1):51-55. doi: 10.1093/ejo/cjab022. PMID 33950232
- [Background] Al-Moghrabi D, Salazar FC, Pandis N, Fleming PS. Compliance with removable orthodontic appliances and adjuncts: A systematic review and meta-analysis. Am J Orthod Dentofacial Orthop. 2017 Jul;152(1):17-32. doi: 10.1016/j.ajodo.2017.03.019. PMID 28651764
- [Background] Al-Moghrabi D, Littlewood SJ, Fleming PS. Orthodontic retention protocols: an evidence-based overview. Br Dent J. 2021 Jun;230(11):770-776. doi: 10.1038/s41415-021-2954-7. Epub 2021 Jun 11. PMID 34117437
- [Background] Thickett E, Power S. A randomized clinical trial of thermoplastic retainer wear. Eur J Orthod. 2010 Feb;32(1):1-5. doi: 10.1093/ejo/cjp061. Epub 2009 Oct 14. PMID 19828592
- [Background] Saub R, Locker D, Allison P. Derivation and validation of the short version of the Malaysian Oral Health Impact Profile. Community Dent Oral Epidemiol. 2005 Oct;33(5):378-83. doi: 10.1111/j.1600-0528.2005.00242.x. PMID 16128798
- [Background] Mohd Tahir N, Wan Hassan WN, Saub R. Comparing retainers constructed on conventional stone models and on 3D printed models: a randomized crossover clinical study. Eur J Orthod. 2019 Aug 8;41(4):370-380. doi: 10.1093/ejo/cjy063. PMID 30321319